CLINICAL TRIAL: NCT03195621
Title: Treatment Strategy for Critical Lesions of Coronary Artery Disease
Brief Title: Critical Treatment of Coronary Artery Disease
Acronym: CTCAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Science and Technology Department of Jiangsu Province (Unknown)
Responsible Party: Principal Investigator, Genshan Ma, Director of cardiology, Southeast University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BE2016785
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease Progression
Keywords: Coronary Artery Disease; Critical lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 2 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional therapy group (Experimental)
  Interventions: Device: Stent implantation
- Conservative treatment group (No Intervention)

INTERVENTIONS:
Device: Stent implantation — Stent placement after risk factors assessment plus FFR or ultrasound or OCT detection for critical lesions.
  Arms: Interventional therapy group

SUMMARY:
Identifying the critical lesion of coronary artery disease and determining the interventional plan are significant for reducing adverse cardiovascular adverse events. The assessment of critical lesion requires the consideration of plaque morphology, tissue composition, and endometrial stress which leading to rupture. In summary, accurate assessment of critical lesions has high application value. In this study, patients with critical coronary artery disease were divided into two groups: an accurate assessment group and a simple assessment group, with the aim to compare the diagnosis and treatment efficiency as well as prognosis, potential cardiovascular risk, possible "excessive" intervention.

ELIGIBILITY:
Inclusion Criteria:

Volunteered to participate in this study and signed an informed consent form;

Men or non-pregnant women ≥ 18 and ≤80 years of age;

Lesion is located in a coronary artery and stenosis is between 50-75%;

Exclusion Criteria:

Severe liver and kidney diseases (GFR<60 ml/min/1.73m2 or CTP≥6 score);

Moderate to severe hypertension (after standard antihypertensive therapy, blood pressure higher than 160/100mmHg);

Patients with hemodynamic or electrical instability (including shock);

Coagulation disorders associated with significant bleeding tendency (eg, hypersensitivity, active bleeding, moderate or severe liver disease, GI bleed within the past 6 months, major surgery within 30 days);

Patients with ischemic stroke within one week;

Any contraindication against the use of anti-platelet drugs such as aspirin;

Platelet count less than 100 x 109/L, haemoglobin (Hb) level less than 100 g/L;

Researchers involved in the study and / or immediate family members;

Participation in another investigation drug or device study in the past 30 days before enrollment;

Involvement in the planning and conduct of the study (applies to staffs at study sites);

Suffering from serious arrhythmias include recurrent ventricular tachycardia or ventricular fibrillation;

Pregnancy or lactation or females of child-bearing potential with the plan of pregnancy in one year;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular adverse events | one year after enrollment
  Cardiac death, myocardial infarction, target vessel revascularization, target lesion revascularization and stent thrombosis

SECONDARY OUTCOMES:
Chest pain | one year after enrollment
  Frequency of angina pectoris

CONTACTS AND LOCATIONS:
Overall Officials: Gen-shan Ma, Ph.D, Study Director — Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
We do not decide whether to share individual participant data